CLINICAL TRIAL: NCT04210635
Title: Evaluation of a Comprehensive Approach in the Management of Anxiety in Intensive Care Unit Including Olfactotherapy
Brief Title: Management of Anxiety in Intensive Care Unit Including Olfactotherapy
Acronym: OCEAN
Status: Completed | Type: Observational
Sponsor: Laboratoires Arkopharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019- A01304-53
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ZEN cart — essential oils + relaxing music + dim light

SUMMARY:
The OCEAN observational study is a pilot study. The aim is to validate the interest of the intervention of essential oils, relaxing music and dim light on the anxiety of patient who are in the intensive care unit.

DETAILED DESCRIPTION:
The primary endpoint is a numeric scale varying from 0 (no anxiety) to 10 (anxiety maximum).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in one of the departments participating in the study
* Presenting moderate to high intensity anxiety (Digital scale ≥ 5);

Exclusion Criteria:

* Having already benefited from the "ZEN cart"
* Having taken an anxiolytic during the past 48 hours
* Patient (s) intubated and / or sedated
* Allergy or known intolerance to one of the essential oils used
* Respiratory allergies, asthma, or a history of seizures
* Unable to understand the information note (linguistic reason, or related to his medical condition)
* Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is made up of adult patients (aged over 18) hospitalized in the intensive care unit and expressing a complaint or presenting a state of anxiety during their hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
measurement of the evolution of anxiety | 6 hours
  The main objective of this study is to measure the evolution of the patient's anxiety between H0 (start of a "ZEN cart" session) and H6 (end of the "ZEN cart" session).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Arnault Tzanck, Saint-Laurent-du-Var, France